CLINICAL TRIAL: NCT04755764
Title: The Effect of Labetalol, Atenolol, and Nifedipine on Maternal Hemodynamics Measured by Impedance Cardiography in Early Pregnancy
Brief Title: Effect of Labetalol, Atenolol, and Nifedipine on Maternal Hemodynamics Measured by ICG in Early Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Jesse Cottrell, Assistant Professor, Marshall University
Other Study IDs: 1681431
Record Dates: First submitted 2021-01-27; First posted 2021-02-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Systolic Hypertension; Pregnancy Related; Diastolic Hypertension; Cardiac Output, Low; Cardiac Output, High
MeSH Terms: conditions — Isolated Systolic Hypertension; Cardiac Output, Low; Cardiac Output, High | interventions — Labetalol; Atenolol; Nifedipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Beta blockade: Beta blocker (labetalol or atenolol) will be given for a cardiac output >8 l/min.
  Interventions: Drug: Labetalol; Drug: Atenolol
- Nifedipine: Nifedipine will be given for a mean arterial pressure >100.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Labetalol — Beta blocker
  Other Names: Normodyne; Trandate
  Groups: Beta blockade
Drug: Atenolol — Beta blocker
  Other Names: Tenormin
  Groups: Beta blockade
Drug: Nifedipine — Calcium channel blocker
  Other Names: Adalat CC; Afeditab CR; Nifediac CC; Nifedical XL; Procardia; Procardia XL
  Groups: Nifedipine

SUMMARY:
The purpose of the research is to characterize the effect of labetalol, atenolol, and nifedipine on maternal hemodynamics early in pregnancy. Patients will be given medication based on their hemodynamics and asked to return for a repeat measurement.

DETAILED DESCRIPTION:
When a patient presents to the Maternal Hypertension Center at Cabell Huntington Hospital, she will receive a non-invasive hemodynamic assessment via the NICaS system as per usual protocol. The NICaS system uses impedance cardiography which provides a reliable assessment of cardiovascular, respiratory, and fluid parameters. In typical practice, the vasodilator nifedipine is initiated for increased systemic vascular resistance and elevated cardiac output is treated with beta blockade (via either atenolol or labetalol). The medication to be given to each subject will be based on their hemodynamics. Specifically, nifedipine will be given for a mean arterial pressure >100 and a beta blocker will be given for a cardiac output >8 l/min. The patients will be asked to return in one week for repeat ICG measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Maternal Hypertension Center at Cabell Huntington Hospital
* English speaking
* 18-45 years old.
* Willing to provide informed consent
* Gestational age prior to 15 weeks gestation

Exclusion Criteria:

* Non-English speaking patients, patients
* <18 years old or >45 years old
* Not willing or able to provide consent
* Gestational age >15 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Patients presenting to the Maternal Hypertension Center at Cabell Huntington Hospital. Consent will be obtained prior to enrollment. Patient age range will be from age 18 to approximately 45.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Initial assessment of hemodynamic parameters will be measured. A change from baseline will be assessed one week later.
  Measured in mmHg
Diastolic blood pressure | Initial assessment of hemodynamic parameters will be measured. A change from baseline will be assessed one week later.
  Measured in mmHg
Mean arterial pressure | Initial assessment of hemodynamic parameters will be measured. A change from baseline will be assessed one week later.
  Measured in mmHg
Heart rate | Initial assessment of hemodynamic parameters will be measured. A change from baseline will be assessed one week later.
  Measured in beats per minute
Cardiac output | Initial assessment of hemodynamic parameters will be measured. A change from baseline will be assessed one week later.
  Measured in liters per minute
Systemic vascular resistance | Initial assessment of hemodynamic parameters will be measured. A change from baseline will be assessed one week later.
  Measured by dynes · sec/cm^-5

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Cottrell, MD, Principal Investigator — Marshall University
Locations (1):
- Maternal Hypertension Center at Cabell Huntington Hospital, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided